CLINICAL TRIAL: NCT02896751
Title: Custom 3-D Printed Noninvasive Ventilation Mask
Brief Title: Use of a 3D Printer to Make Custom Sleep Masks for Positive Airway Pressure Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIN001-3D Printer NIV Mask
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2023-08

CONDITIONS: Sleep Apnea; Pediatric Sleep Apnea
Keywords: CPAP; Noninvasive Ventilation Mask
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3D Printed NIV Mask (Experimental): 3D imaging and use of a custom mask from 3D printer
  Interventions: Device: 3D printed NIV mask

INTERVENTIONS:
Device: 3D printed NIV mask — use of 3D printed mask

SUMMARY:
This is a small pilot study to look at the feasibility of creating a customized sleep mask for use with Continuous Positive Airway Pressure (CPAP) or other similar treatments for sleep apnea. The participant will have three dimensional (3D) pictures of the face taken by special cameras. The pictures will be sent to a 3D printer and a mask will be created based on the participant's face contours. The participant will use the mask for about 6 months. The study will measure the amount it is used during sleep and if there is an increase in reported comfort.

DETAILED DESCRIPTION:
The aim of this study is to improve adherence and effectiveness of noninvasive ventilation by decreasing the side effects commonly seen with noninvasive ventilation. Studies have shown that even though noninvasive ventilation (NIV) with positive airway pressure (PAP) is successful at treating obstructive sleep apnea and hypoventilation, individuals have poor compliance with therapy. The reasons for poor compliance are numerous, but one significant and continually reported reason is poor mask fit. A poor mask fit is not only uncomfortable, but frequently causes side effects such as dry eyes, congestion, skin irritation and breakdown, and ineffective ventilation from inadequate pressures due to air leaking around the mask. Pediatric patients tend to be especially difficult to fit with conventional masks because of their smaller facial features and the lack of masks developed for pediatric use.

In this study, patients will be fitted with a custom made NIV mask following facial imaging with a 3D camera (Artec 3D Scanner). The facial image will be used to construct an NIV mask model using computer design software that will then be created by using a 3D printer.

ELIGIBILITY:
Inclusion Criteria:

* On stable NIV settings for a minimum of 2 months.

Exclusion Criteria:

* New diagnosis

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
CPAP Adherence | 6 months
  Measure CPAP usage

CONTACTS AND LOCATIONS:
Overall Officials: Narong Simakajornboon, MD, Principal Investigator — Cincinnati Children's Hopital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with treating sleep physicians to improve care
Supporting Information: CSR
Time Frame: Data will be shared with treating sleep physicians to improve care
Access Criteria: Data will be shared with treating sleep physicians to improve care

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT02896751/Prot_SAP_000.pdf